CLINICAL TRIAL: NCT03978637
Title: An Open-Label, Single-Arm, Phase 1/2 Study Evaluating the Safety and Efficacy of Itacitinib in Participants With Bronchiolitis Obliterans Syndrome Following Lung Transplantation
Brief Title: Safety and Efficacy of Itacitinib in Participants With Bronchiolitis Obliterans Syndrome Following Lung Transplantation
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Business Decision
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: INCB 39110-214; 2019-004171-39 (EudraCT Number)
Record Dates: First submitted 2019-06-05; First posted 2019-06-07 (Actual); Results first posted 2025-01-29 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Bronchiolitis Obliterans Syndrome
Keywords: Bronchiolitis obliterans syndrome; lung transplant; JAK1 inhibitor
MeSH Terms: conditions — Bronchiolitis Obliterans Syndrome | interventions — itacitinib; INCB039110

STUDY DESIGN:
Intervention Model Description: Phase 1 Itacitinib administered orally followed by phase 2; Itacitinib administered orally at the recommended dose from Phase 1.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Itacitinib 300 mg (Experimental): Phase 1: Itacitinib 300 mg twice daily. There can be required dose adjustments in the protocol for concurrent CYP3A administration.
  Interventions: Drug: Itacitinib
- Itacitinib 400 mg (Experimental): Phase 1: Itacitinib 400 mg once daily. There can be required dose adjustments in the protocol for concurrent CYP3A administration.
  Interventions: Drug: Itacitinib
- Itacitinib 600 mg (Experimental): Phase 1: Itacitinib 600 mg once daily. There can be required dose adjustments in the protocol for concurrent CYP3A administration
  Interventions: Drug: Itacitinib
- Itacitinib (Experimental): Phase 2: Itacitinib administered orally at the recommended dose from Phase 1.
  Interventions: Drug: Itacitinib

INTERVENTIONS:
Drug: Itacitinib — Itacitinib administered orally at the specified dose.
  Other Names: INCB039110

SUMMARY:
The purpose of this study is to evaluate the safety, efficacy, pharmacokinetics, and pharmacodynamics of itacitinib in participants with post-lung transplant bronchiolitis obliterans syndrome (BOS).

ELIGIBILITY:
Inclusion Criteria:

* Double lung transplantation ≥ 1 year before informed consent. Confirmed BOS progression to Grade 1, 2, or 3 diagnosed within 1 year of screening

  *Confirmed BOS progression to Grade 1, 2, or 3 diagnosed within 2 years of screening AND:
* A ≥ 200 mL decrease in FEV1 in the previous 12 months

OR

*A ≥ 50 mL decrease in FEV1 in the last 2 measurements.

• Willingness to avoid pregnancy or fathering children.

Exclusion Criteria:

* History of a single lung transplant
* FEV1 decline attributable to cause(s) other than BOS.
* Participants who have had any significant change (eg, addition of new agents) in an immunosuppressive regimen in the 4 weeks before screening.
* Untreated and/or symptomatic gastroesophageal reflux disease.
* Significant infectious comorbidities including invasive fungal disease, B. Cepacia, non TB mycobacteria, or TB.
* Receipt of JAK inhibitor therapy after lung transplant for any indication. Treatment with a JAK inhibitor before lung transplant is permitted.
* Laboratory values at screening outside the protocol-defined ranges.
* Active HBV or HCV infection that requires treatment, or at risk for HBV reactivation (ie, positive HBsAg).
* Known HIV infection.
* History of active malignancy within 3 years of screening.
* Women who are pregnant or breastfeeding.
* Treatment with an investigational agent, procedure, or device within 30 days of enrollment, or within 5 half-lives of the investigational product, whichever is longer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2020-02-04 (Actual); Primary Completion 2023-10-13 (Actual); Study Completion 2023-10-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin O'Hayer, MD, Study Director — Incyte Corporation
Locations (9):
- United States (7):
  - University of California, Los Angeles - David Geffen School of Medicine, Los Angeles, California
  - Brigham and Women'S Faulkner Hospitals Inc, Boston, Massachusetts
  - Duke University Health System, Durham, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Temple University Department of Thoracic Medicine and Surgery, Philadelphia, Pennsylvania
  - UPMC, Pittsburgh, Pennsylvania
- Universitaire Ziekenhuis Leuven - Gasthuisberg, Leuven, Belgium
- University Health Network Toronto General Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study was conducted at 7 study centers in the United States, Canada, and Belgium. The site in Canada had a screen failure but did not recruit any participants.
Groups:
- Itacitinib 300/200 mg: Participants not taking a concomitant strong CYP3A inhibitor received a starting dose of itacitinib 300 milligrams (mg) twice daily (BID). Participants taking a concomitant strong CYP3A inhibitor received a starting dose of itacitinib 200 mg BID. Participants may have had dose reductions or modifications during the course of treatment based on adverse events, clinical evaluation, changes to concomitant medications, and laboratory assessments. Itacitinib treatment was continued until progression of bronchiolitis obliterans syndrome (defined as a ≥10% absolute decrease from Baseline in forced expiratory volume in 1 second (FEV1), confirmed by 2 consecutive spirometric assessments ≥3 weeks apart), unacceptable toxicity, loss of clinical benefit, or withdrawal of consent.
- Itacitinib 400/300 mg: Participants not taking a concomitant strong CYP3A inhibitor received a starting dose of itacitinib 400 mg once daily (QD). Participants taking a concomitant strong CYP3A inhibitor received a starting dose of itacitinib 300 mg QD. Participants may have had dose reductions or modifications during the course of treatment based on adverse events, clinical evaluation, changes to concomitant medications, and laboratory assessments. Itacitinib treatment was continued until progression of bronchiolitis obliterans syndrome (defined as a ≥10% absolute decrease from Baseline in FEV1, confirmed by 2 consecutive spirometric assessments ≥3 weeks apart), unacceptable toxicity, loss of clinical benefit, or withdrawal of consent.
- Itacitinib 600/400 mg: Participants not taking a concomitant strong CYP3A inhibitor received a starting dose of itacitinib 600 mg QD. Participants taking a concomitant strong CYP3A inhibitor received a starting dose of itacitinib 400 mg QD. Participants may have had dose reductions or modifications during the course of treatment based on adverse events, clinical evaluation, changes to concomitant medications, and laboratory assessments. Itacitinib treatment was continued until progression of bronchiolitis obliterans syndrome (defined as a ≥10% absolute decrease from Baseline in FEV1, confirmed by 2 consecutive spirometric assessments ≥3 weeks apart), unacceptable toxicity, loss of clinical benefit, or withdrawal of consent.
- Other: Participants received a starting dose of itacitinib 200 mg QD. Participants may have had dose reductions or modifications during the course of treatment based on adverse events, clinical evaluation, changes to concomitant medications, and laboratory assessments. Itacitinib treatment was continued until progression of bronchiolitis obliterans syndrome (defined as a ≥10% absolute decrease from Baseline in FEV1, confirmed by 2 consecutive spirometric assessments ≥3 weeks apart), unacceptable toxicity, loss of clinical benefit, or withdrawal of consent.
Period: Overall Study
Arm/Group | Itacitinib 300/200 mg | Itacitinib 400/300 mg | Itacitinib 600/400 mg | Other
Started | 7 | 7 | 8 | 1
Completed | 6 | 2 | 3 | 1
Not Completed | 1 | 5 | 5 | 0
Not completed — Death | 0 | 2 | 2 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0
Not completed — Transitioned to Itacitinib Rollover Trial | 1 | 3 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Itacitinib 300/200 mg | Itacitinib 400/300 mg | Itacitinib 600/400 mg | Other | Total
Number analyzed (Participants) | 7 | 7 | 8 | 1 | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 5 | 5 | 6 | 1 | 17
  >=65 years | 2 | 2 | 2 | 0 | 6
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 2 | 2 | 1 | 1 | 6
  Male | 5 | 5 | 7 | 0 | 17
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White/Caucasian | 6 | 6 | 7 | 1 | 20
  Black/African-American | 1 | 1 | 1 | 0 | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 0 | 1
  Not Hispanic or Latino | 6 | 7 | 7 | 1 | 21
  Unknown | 0 | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Any Treatment-emergent Adverse Event (TEAE)
Description: An adverse event (AE) was defined as any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug-related. An AE could therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of study treatment. A TEAE was defined as either an AE reported for the first time or the worsening of a pre-existing condition after the first dose of itacitinib until 30 days after the last dose of itacitinib.
Time Frame: up to approximately 162 weeks
Population: Full Analysis Set: all participants enrolled in the study who received at least 1 dose of itacitinib
Measure: Count of Participants; unit: Participants
Arm/Group | Itacitinib 300/200 mg | Itacitinib 400/300 mg | Itacitinib 600/400 mg | Other
Number analyzed (Participants) | 7 | 7 | 8 | 1
Participants | 7 | 7 | 8 | 1

2. Primary Outcome: Number of Participants With Any Grade 3 or Higher TEAE
Description: An AE was defined as any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug-related. A TEAE was defined as either an AE reported for the first time or the worsening of a pre-existing condition after the first dose of itacitinib until 30 days after the last dose of itacitinib. The severity of AEs was assessed using Common Terminology Criteria for Adverse Events v5.0. Grade 1: mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; treatment not indicated. Grade 2: moderate; minimal, local, or noninvasive treatment indicated; limiting age appropriate activities of daily living. Grade 3: severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self-care activities of daily living. Grade 4: life-threatening consequences; urgent treatment indicated. Grade 5: fatal.
Time Frame: up to approximately 162 weeks
Population: Full Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Itacitinib 300/200 mg | Itacitinib 400/300 mg | Itacitinib 600/400 mg | Other
Number analyzed (Participants) | 7 | 7 | 8 | 1
Participants | 6 | 7 | 6 | 1

3. Primary Outcome: Change From Baseline in Forced Expiratory Volume in 1 Second (FEV1) at Week 12
Description: FEV1 was defined as the volume of air exhaled in 1 second. Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Baseline; Week 12
Population: Full Analysis Set. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | Itacitinib 300/200 mg | Itacitinib 400/300 mg | Itacitinib 600/400 mg | Other
Number analyzed (Participants) | 7 | 7 | 8 | 1
liters
  Baseline | 1.72 (0.962) | 1.57 (0.672) | 1.59 (0.511) | 1.34 (NA) — Standard deviation cannot be reported for a single participant.
  Change from Baseline: number analyzed (Participants) | 5 | 7 | 5 | 0
  Change from Baseline | 0.09 (0.168) | 0.04 (0.114) | 0.22 (0.571) |

4. Primary Outcome: Phase 2: FEV1 Response Rate
Description: FEV1 response rate was defined as the percentage of participants demonstrating a ≥10% absolute increase in FEV1 compared with Baseline, confirmed by 2 consecutive spirometric assessments ≥1 week apart.
Time Frame: Baseline through Week 12
Population: A business decision was made to terminate the study before the initiation of Part 2. The decision to terminate the study was unrelated to safety concerns.
Groups:
- Recommended Phase 2 Dose (RP2D): Participants were to receive itacitinib at the RP2D. Itacitinib treatment was to be continued until progression of bronchiolitis obliterans syndrome (defined as a ≥10% absolute decrease from Baseline in FEV1, confirmed by 2 consecutive spirometric assessments ≥3 weeks apart), unacceptable toxicity, loss of clinical benefit, or withdrawal of consent.
Arm/Group | Recommended Phase 2 Dose (RP2D)
Number analyzed (Participants) | 0

5. Secondary Outcome: Phase 1: Duration of FEV1 Response
Description: Duration of FEV1 response was defined as the interval between the onset of response and the earliest of bronchiolitis obliterans syndrome (BOS) progression, loss of clinical benefit as determined by the investigator, or death.
Time Frame: up to 34.9 months
Population: Full Analysis Set. Only those participants with a response were analyzed.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Itacitinib 300/200 mg | Itacitinib 400/300 mg | Itacitinib 600/400 mg | Other
Number analyzed (Participants) | 1 | 2 | 1 | 0
days | NA [NA to NA] — The median and the upper and lower limits of the confidence interval were not estimable because there were too few events of BOS progression or loss of clinical benefit. | 491.5 [401.0 to NA] — The upper limit of the confidence interval was not estimable because there were too few events of BOS progression or loss of clinical benefit. | NA [NA to NA] — The median and the upper and lower limits of the confidence interval were not estimable because there were too few events of BOS progression or loss of clinical benefit. |

6. Secondary Outcome: Phase 2: Duration of FEV1 Response
Description: Duration of FEV1 response was defined as the interval between the onset of response and the earliest of bronchiolitis obliterans syndrome progression, loss of clinical benefit as determined by the investigator, or death.
Time Frame: up to 24 months
Population: as for outcome 4
Arm/Group | Recommended Phase 2 Dose (RP2D)
Number analyzed (Participants) | 0

7. Secondary Outcome: Phase 1: Time to Progression
Description: Time to progression was defined as defined as the interval between the start of treatment and bronchiolitis obliterans syndrome progression (≥10% absolute decrease in FEV1 compared to baseline), or death.
Time Frame: up to 36.4 months
Population: Full Analysis Set
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Itacitinib 300/200 mg | Itacitinib 400/300 mg | Itacitinib 600/400 mg | Other
Number analyzed (Participants) | 7 | 7 | 8 | 1
days | 516.0 [13.0 to NA] — The upper limit of the confidence interval was not estimable because too few participants had disease progression or died. | 485.0 [19.0 to 750.0] | NA [56.0 to NA] — The median and the upper limit of the confidence interval were not estimable because too few participants had disease progression or died. | NA [NA to NA] — The median and the upper and lower limits of the confidence interval were not estimable because too few participants had disease progression or died.

8. Secondary Outcome: Phase 2: Time to Progression
Description: as for outcome 7
Time Frame: up to 24 months
Population: as for outcome 4
Arm/Group | Recommended Phase 2 Dose (RP2D)
Number analyzed (Participants) | 0

9. Secondary Outcome: Phase 1: Change From Baseline in the St. George's Respiratory Questionnaire (SGRQ) Total Score
Description: The SGRQ is a disease-specific instrument designed to measure the impact on overall health, daily life, and perceived well-being in participants with obstructive airway disease. It consists of 50 items covering 3 domains: symptoms (8 items), activity (16 items), and impacts (26 items). A component score is calculated for each of the 3 domains. One total score is calculated if none of the component scores is missing. All scales (both domain and total) have a score ranging between 0 and 100, with higher scores indicating a worse quality of life. Change from (CFB) Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Baseline; up to 158.4 weeks
Population: Full Analysis Set. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Itacitinib 300/200 mg | Itacitinib 400/300 mg | Itacitinib 600/400 mg | Other
Number analyzed (Participants) | 7 | 7 | 8 | 1
scores on a scale
  Baseline | 51.21 (16.740) | 38.79 (15.165) | 52.94 (20.961) | 19.86 (NA) — Standard deviation cannot be reported for a single participant.
  Change from Baseline at Week 12: number analyzed (Participants) | 5 | 7 | 5 | 1
  Change from Baseline at Week 12 | -5.70 (8.792) | -4.55 (7.627) | 0.87 (15.895) | -1.84 (NA) — Standard deviation cannot be reported for a single participant.
  Change from Baseline at End of Treatment: number analyzed (Participants) | 1 | 2 | 0 | 1
  Change from Baseline at End of Treatment | 13.17 (NA) — Standard deviation cannot be reported for a single participant. | 6.82 (3.416) |  | -2.34 (NA) — Standard deviation cannot be reported for a single participant.

10. Secondary Outcome: Phase 2: Change From Baseline in the SGRQ Total Score
Description: The SGRQ is a disease-specific instrument designed to measure the impact on overall health, daily life, and perceived well-being in participants with obstructive airway disease. It consists of 50 items covering 3 domains: symptoms (8 items), activity (16 items), and impacts (26 items). A component score is calculated for each of the 3 domains. One total score is calculated if none of the component scores is missing. All scales (both domain and total) have a score ranging between 0 and 100, with higher scores indicating a worse quality of life. Change from Baseline was to be calculated as the post-Baseline value minus the Baseline value.
Time Frame: up to 24 months
Population: as for outcome 4
Arm/Group | Recommended Phase 2 Dose (RP2D)
Number analyzed (Participants) | 0

11. Secondary Outcome: Phase 1: Change From Baseline in the Quality of Life-Short Form-12 (QOL-SF-12) Questionnaire Scores
Description: The QOL-SF-12 v2 is a 12-item subset of the QOL-SF-36 v2 scale that assesses 8 health concepts related to limitations in physical activities, social activities (SA), bodily pain, general mental and physical health, and vitality. Participants answered each question by selecting pre-specified choices. Score ranges are specified for each item; higher scores indicate better health. Assessment of health score: poor (1) to excellent (5). Moderate activities and climbing stairs score: limited a lot (1) to not limited at all (3). Accomplished less because of physical health (PH) or emotional problems (EP)/limited in work/did work less carefully score: all of the time (1) to none of the time (5). Pain interfered with work score: extremely (1) to not at all (5). Felt calm/peaceful, had a lot of energy, felt depressed, PH or EP interfered with SA score: none of the time (1) to all of the time (6). Change from Baseline (BL) was calculated as the post-BL value minus the BL value.
Time Frame: Baseline; up to 158.4 weeks
Population: Full Analysis Set. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Itacitinib 300/200 mg | Itacitinib 400/300 mg | Itacitinib 600/400 mg | Other
Number analyzed (Participants) | 7 | 7 | 8 | 1
scores on a scale
  Baseline, assessment of health | 2.60 (0.748) | 2.80 (0.748) | 2.53 (1.100) | 3.40 (NA) — Standard deviation cannot be reported for a single participant.
  Change from Baseline (CFB) at Week 12, assessment of health: number analyzed (Participants) | 5 | 7 | 5 | 1
  Change from Baseline (CFB) at Week 12, assessment of health | -0.28 (0.626) | 0.14 (0.378) | -0.20 (0.447) | 0.00 (NA) — Standard deviation cannot be reported for a single participant.
  CFB at end of treatment (EOT), assessment of health: number analyzed (Participants) | 1 | 2 | 1 | 1
  CFB at end of treatment (EOT), assessment of health | 0.00 (NA) — Standard deviation cannot be reported for a single participant. | -0.70 (0.990) | 0.00 (NA) — Standard deviation cannot be reported for a single participant. | 0.00 (NA) — Standard deviation cannot be reported for a single participant.
  Baseline, Moderate Activities: number analyzed (Participants) | 6 | 7 | 8 | 1
  Baseline, Moderate Activities | 1.50 (0.837) | 2.00 (0.577) | 1.50 (0.756) | 2.00 (NA) — Standard deviation cannot be reported for a single participant.
  CFB at Week 12, Moderate Activities: number analyzed (Participants) | 5 | 7 | 5 | 1
  CFB at Week 12, Moderate Activities | 0.20 (0.447) | 0.00 (0.577) | 0.20 (0.447) | 1.00 (NA) — Standard deviation cannot be reported for a single participant.
  CFB at EOT, Moderate Activities: number analyzed (Participants) | 0 | 2 | 0 | 1
  CFB at EOT, Moderate Activities |  | -0.50 (0.707) |  | 0.00 (NA) — Standard deviation cannot be reported for a single participant.
  Baseline, Climbing Several Flights of Stairs: number analyzed (Participants) | 6 | 7 | 8 | 1
  Baseline, Climbing Several Flights of Stairs | 1.33 (0.816) | 1.86 (0.690) | 1.38 (0.518) | 2.00 (NA) — Standard deviation cannot be reported for a single participant.
  CFB at Week 12, Climbing Several Flights of Stairs: number analyzed (Participants) | 5 | 7 | 5 | 1
  CFB at Week 12, Climbing Several Flights of Stairs | 0.20 (0.837) | 0.00 (0.577) | 0.00 (0.000) | 0.00 (NA) — Standard deviation cannot be reported for a single participant.
  CFB at Week EOT, Climbing Several Flights of Stairs: number analyzed (Participants) | 0 | 2 | 0 | 1
  CFB at Week EOT, Climbing Several Flights of Stairs |  | -1.00 (0.000) |  | 0.00 (NA) — Standard deviation cannot be reported for a single participant.
  Baseline, Accomplished Less than Liked because of Physical Health | 2.14 (0.900) | 3.14 (1.345) | 2.63 (1.302) | 4.00 (NA) — Standard deviation cannot be reported for a single participant.
  CFB at Week 12, Accomplished Less than Liked because of Physical Health: number analyzed (Participants) | 5 | 7 | 5 | 1
  CFB at Week 12, Accomplished Less than Liked because of Physical Health | 0.20 (1.095) | 0.14 (1.773) | -0.80 (0.837) | 1.00 (NA) — Standard deviation cannot be reported for a single participant.
  CFB at EOT, Accomplished Less than Liked because of Physical Health: number analyzed (Participants) | 1 | 2 | 0 | 1
  CFB at EOT, Accomplished Less than Liked because of Physical Health | -1.00 | -0.50 (3.536) |  | 1.00 (NA) — Standard deviation cannot be reported for a single participant.
  Baseline, Limited in Work/Other Activities | 2.14 (0.900) | 2.86 (0.900) | 2.50 (1.309) | 4.00 (NA) — Standard deviation cannot be reported for a single participant.
  CFB at Week 12, Limited in Work/Other Activities: number analyzed (Participants) | 5 | 7 | 5 | 1
  CFB at Week 12, Limited in Work/Other Activities | -0.20 (0.447) | 0.43 (0.787) | -0.40 (1.140) | 0.00 (NA) — Standard deviation cannot be reported for a single participant.
  CFB at EOT, Limited in Work/Other Activities: number analyzed (Participants) | 1 | 2 | 0 | 1
  CFB at EOT, Limited in Work/Other Activities | -1.00 (NA) — Standard deviation cannot be reported for a single participant. | 0.50 (0.707) |  | 0.00 (NA) — Standard deviation cannot be reported for a single participant.
  Baseline, Accomplished Less than Liked because of Emotional Problems | 4.14 (0.900) | 3.57 (0.976) | 4.13 (1.246) | 5.00 (NA) — Standard deviation cannot be reported for a single participant.
  CFB at Week 12, Accomplished Less than Liked because of Emotional Problems: number analyzed (Participants) | 5 | 7 | 5 | 1
  CFB at Week 12, Accomplished Less than Liked because of Emotional Problems | 0.20 (1.095) | 0.00 (1.291) | -0.20 (1.483) | 0.00 (NA) — Standard deviation cannot be reported for a single participant.
  CFB at EOT, Accomplished Less than Liked because of Emotional Problems: number analyzed (Participants) | 1 | 2 | 0 | 1
  CFB at EOT, Accomplished Less than Liked because of Emotional Problems | 1.00 (NA) — Standard deviation cannot be reported for a single participant. | -2.00 (1.414) |  | 0.00 (NA) — Standard deviation cannot be reported for a single participant.
  Baseline, Did Work/Activities Less Carefully | 4.14 (0.900) | 3.71 (0.756) | 4.25 (1.035) | 5.00 (NA) — Standard deviation cannot be reported for a single participant.
  CFB at Week 12, Did Work/Activities Less Carefully: number analyzed (Participants) | 5 | 7 | 5 | 1
  CFB at Week 12, Did Work/Activities Less Carefully | 0.20 (1.095) | -0.29 (1.380) | -0.80 (1.095) | 0.00 (NA) — Standard deviation cannot be reported for a single participant.
  CFB at EOT, Did Work/Activities Less Carefully: number analyzed (Participants) | 1 | 2 | 0 | 1
  CFB at EOT, Did Work/Activities Less Carefully | 1.00 (NA) — Standard deviation cannot be reported for a single participant. | -2.00 (0.000) |  | 0.00 (NA) — Standard deviation cannot be reported for a single participant.
  Baseline, Pain Interfered with Normal Work | 4.29 (1.254) | 4.00 (0.816) | 4.00 (1.309) | 5.00 (NA) — Standard deviation cannot be reported for a single participant.
  CFB at Week 12, Pain Interfered with Normal Work: number analyzed (Participants) | 5 | 7 | 5 | 1
  CFB at Week 12, Pain Interfered with Normal Work | 0.00 (0.707) | 0.14 (1.215) | -0.20 (1.095) | 0.00 (NA) — Standard deviation cannot be reported for a single participant.
  CFB at EOT, Pain Interfered with Normal Work: number analyzed (Participants) | 1 | 2 | 0 | 1
  CFB at EOT, Pain Interfered with Normal Work | -1.00 (NA) — Standard deviation cannot be reported for a single participant. | 0.00 (0.000) |  | 0.00 (NA) — Standard deviation cannot be reported for a single participant.
  Baseline, Felt Calm/Peaceful | 3.86 (0.378) | 3.14 (0.690) | 3.50 (1.195) | 5.00 (NA) — Standard deviation cannot be reported for a single participant.
  CFB at Week 12, Felt Calm/Peaceful: number analyzed (Participants) | 5 | 7 | 5 | 1
  CFB at Week 12, Felt Calm/Peaceful | -0.20 (1.643) | 0.29 (1.113) | -0.20 (1.095) | 0.00 (NA) — Standard deviation cannot be reported for a single participant.
  CFB at EOT, Felt Calm/Peaceful: number analyzed (Participants) | 1 | 2 | 0 | 1
  CFB at EOT, Felt Calm/Peaceful | 0.00 (NA) — Standard deviation cannot be reported for a single participant. | -1.00 (1.414) |  | 0.00 (NA) — Standard deviation cannot be reported for a single participant.
  Baseline, Had a Lot of Energy | 2.29 (1.113) | 2.71 (0.756) | 2.25 (0.886) | 4.00 (NA) — Standard deviation cannot be reported for a single participant.
  CFB at Week 12, Had a Lot of Energy: number analyzed (Participants) | 5 | 7 | 5 | 1
  CFB at Week 12, Had a Lot of Energy | 0.00 (0.707) | 0.43 (1.512) | -0.60 (1.140) | 0.00 (NA) — Standard deviation cannot be reported for a single participant.
  CFB at EOT, Had a Lot of Energy: number analyzed (Participants) | 1 | 2 | 0 | 1
  CFB at EOT, Had a Lot of Energy | 0.00 (NA) — Standard deviation cannot be reported for a single participant. | -1.00 (0.000) |  | 1.00 (NA) — Standard deviation cannot be reported for a single participant.
  Baseline, Felt Downhearted/Depressed | 4.43 (0.787) | 3.14 (0.690) | 4.75 (0.463) | 5.00 (NA) — Standard deviation cannot be reported for a single participant.
  CFB at Week 12, Felt Downhearted/Depressed: number analyzed (Participants) | 5 | 7 | 5 | 1
  CFB at Week 12, Felt Downhearted/Depressed | -0.20 (0.447) | 0.43 (0.787) | -0.80 (1.304) | 0.00 (NA) — Standard deviation cannot be reported for a single participant.
  CFB at EOT, Felt Downhearted/Depressed: number analyzed (Participants) | 1 | 2 | 0 | 1
  CFB at EOT, Felt Downhearted/Depressed | 1.00 (NA) — Standard deviation cannot be reported for a single participant. | -0.50 (0.707) |  | 0.00 (NA) — Standard deviation cannot be reported for a single participant.
  Baseline, Interference with Social Activity | 4.43 (0.787) | 4.14 (0.900) | 2.75 (1.581) | 5.00 (NA) — Standard deviation cannot be reported for a single participant.
  CFB at Week 12, Interference with Social Activity: number analyzed (Participants) | 5 | 7 | 5 | 1
  CFB at Week 12, Interference with Social Activity | -0.20 (0.447) | -0.29 (1.380) | 0.00 (1.581) | 0.00 (NA) — Standard deviation cannot be reported for a single participant.
  CFB at EOT, Interference with Social Activity: number analyzed (Participants) | 1 | 2 | 0 | 1
  CFB at EOT, Interference with Social Activity | 1.00 (NA) — Standard deviation cannot be reported for a single participant. | -1.00 (1.414) |  | 0.00 (NA) — Standard deviation cannot be reported for a single participant.

12. Secondary Outcome: Phase 2: Change From Baseline in QOL-SF-12 Questionnaire Scores
Description: The QOL-SF-12 v2 is a 12-item subset of the QOL-SF-36 v2 scale that assesses 8 health concepts related to limitations in physical activities, social activities (SA), bodily pain, general mental and physical health, and vitality. Participants answered each question by selecting pre-specified choices. Score ranges are specified for each item; higher scores indicate better health. Assessment of health score: poor (1) to excellent (5). Moderate activities and climbing stairs score: limited a lot (1) to not limited at all (3). Accomplished less because of physical health (PH) or emotional problems (EP)/limited in work/did work less carefully score: all of the time (1) to none of the time (5). Pain interfered with work score: extremely (1) to not at all (5). Felt calm/peaceful, had a lot of energy, felt depressed, PH or EP interfered with SA score: none of the time (1) to all of the time (6). Change from Baseline (BL) was to be calculated as the post-BL value minus the BL value.
Time Frame: up to 24 months
Population: as for outcome 4
Arm/Group | Recommended Phase 2 Dose (RP2D)
Number analyzed (Participants) | 0

13. Secondary Outcome: Phase 1: Number of Participants With the Indicated Responses on the EQ-5D-3L Questionnaire Regarding Their Health State
Description: The EQ-5D-3L essentially consists of 2 components: the EQ-5D descriptive scale and the EQ-VAS. The EQ-5D-3L descriptive system comprises the following 5 dimensions: mobility, self-care, usual activities, anxiety/depression, and pain/discomfort. Each dimension has 3 levels: no problems, some problems, and extreme problems. At each specific visit (starting on Day 1), the participant was asked to indicate their health state. BL=Baseline; EOT=end of treatment.
Time Frame: Baseline; up to 158.4 weeks
Population: Full Analysis Set. Only participants with available data were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Itacitinib 300/200 mg | Itacitinib 400/300 mg | Itacitinib 600/400 mg | Other
Number analyzed (Participants) | 7 | 7 | 8 | 1
Participants
  Mobility, no problems walking about at BL | 1 | 2 | 4 | 1
  Mobility, some problems walking about at BL | 6 | 5 | 4 | 0
  Mobility, confined to bed at BL | 0 | 0 | 0 | 0
  Mobility, no problems walking about at Week 12: number analyzed (Participants) | 5 | 6 | 5 | 1
  Mobility, no problems walking about at Week 12 | 3 | 2 | 3 | 1
  Mobility, some problems walking about at Week 12: number analyzed (Participants) | 5 | 6 | 5 | 1
  Mobility, some problems walking about at Week 12 | 2 | 4 | 2 | 0
  Mobility, confined to bed at Week 12: number analyzed (Participants) | 5 | 6 | 5 | 1
  Mobility, confined to bed at Week 12 | 0 | 0 | 0 | 0
  Mobility, no problems walking about at EOT: number analyzed (Participants) | 0 | 1 | 0 | 1
  Mobility, no problems walking about at EOT | 0 | 0 | 0 | 1
  Mobility, some problems walking about at EOT: number analyzed (Participants) | 0 | 1 | 0 | 1
  Mobility, some problems walking about at EOT | 0 | 1 | 0 | 0
  Mobility, confined to bed at EOT: number analyzed (Participants) | 0 | 1 | 0 | 1
  Mobility, confined to bed at EOT | 0 | 0 | 0 | 0
  Self-care, no problems at BL | 4 | 5 | 6 | 1
  Self-care, some problems at BL | 3 | 2 | 2 | 0
  Self-care, unable to wash or dress self at BL | 0 | 0 | 0 | 0
  Self-care, no problems at Week 12: number analyzed (Participants) | 5 | 6 | 5 | 1
  Self-care, no problems at Week 12 | 4 | 4 | 4 | 1
  Self-care, some problems at Week 12: number analyzed (Participants) | 5 | 6 | 5 | 1
  Self-care, some problems at Week 12 | 0 | 2 | 1 | 0
  Self-care, unable to wash or dress self at Week 12: number analyzed (Participants) | 5 | 6 | 5 | 1
  Self-care, unable to wash or dress self at Week 12 | 1 | 0 | 0 | 0
  Self-care, no problems at EOT: number analyzed (Participants) | 0 | 1 | 0 | 1
  Self-care, no problems at EOT | 0 | 0 | 0 | 1
  Self-care, some problems at EOT: number analyzed (Participants) | 0 | 1 | 0 | 1
  Self-care, some problems at EOT | 0 | 1 | 0 | 0
  Self-care, unable to wash or dress self at EOT: number analyzed (Participants) | 0 | 1 | 0 | 1
  Self-care, unable to wash or dress self at EOT | 0 | 0 | 0 | 0
  Usual activities, no problems at BL | 2 | 3 | 2 | 1
  Usual activities, some problems at BL | 4 | 4 | 5 | 0
  Usual activities, unable to perform usual activities at BL | 1 | 0 | 1 | 0
  Usual activities, no problems at Week 12: number analyzed (Participants) | 5 | 6 | 5 | 1
  Usual activities, no problems at Week 12 | 1 | 2 | 1 | 1
  Usual activities, some problems at Week 12: number analyzed (Participants) | 5 | 6 | 5 | 1
  Usual activities, some problems at Week 12 | 3 | 3 | 3 | 0
  Usual activities, unable to perform usual activities at Week 12: number analyzed (Participants) | 5 | 6 | 5 | 1
  Usual activities, unable to perform usual activities at Week 12 | 1 | 1 | 1 | 0
  Usual activities, no problems at EOT: number analyzed (Participants) | 0 | 1 | 0 | 1
  Usual activities, no problems at EOT | 0 | 0 | 0 | 1
  Usual activities, some problems at EOT: number analyzed (Participants) | 0 | 1 | 0 | 1
  Usual activities, some problems at EOT | 0 | 1 | 0 | 0
  Usual activities, unable to perform usual activities at EOT: number analyzed (Participants) | 0 | 1 | 0 | 1
  Usual activities, unable to perform usual activities at EOT | 0 | 0 | 0 | 0
  Pain/discomfort, no pain/discomfort at BL | 3 | 1 | 4 | 1
  Pain/discomfort, moderate pain/discomfort at BL | 3 | 6 | 4 | 0
  Pain/discomfort, extreme pain/discomfort at BL | 1 | 0 | 0 | 0
  Pain/discomfort, no pain/discomfort at Week 12: number analyzed (Participants) | 5 | 6 | 5 | 1
  Pain/discomfort, no pain/discomfort at Week 12 | 2 | 2 | 2 | 1
  Pain/discomfort, moderate pain/discomfort at Week 12: number analyzed (Participants) | 5 | 6 | 5 | 1
  Pain/discomfort, moderate pain/discomfort at Week 12 | 3 | 4 | 3 | 0
  Pain/discomfort, extreme pain/discomfort at Week 12: number analyzed (Participants) | 5 | 6 | 5 | 1
  Pain/discomfort, extreme pain/discomfort at Week 12 | 0 | 0 | 0 | 0
  Pain/discomfort, no pain/discomfort at EOT: number analyzed (Participants) | 0 | 1 | 0 | 1
  Pain/discomfort, no pain/discomfort at EOT | 0 | 0 | 0 | 1
  Pain/discomfort, moderate pain/discomfort at EOT: number analyzed (Participants) | 0 | 1 | 0 | 1
  Pain/discomfort, moderate pain/discomfort at EOT | 0 | 1 | 0 | 0
  Pain/discomfort, extreme pain/discomfort at EOT: number analyzed (Participants) | 0 | 1 | 0 | 1
  Pain/discomfort, extreme pain/discomfort at EOT | 0 | 0 | 0 | 0
  Anxiety/depression, not anxious/depressed at BL | 6 | 2 | 6 | 1
  Anxiety/depression, moderately anxious/depressed at BL | 1 | 5 | 1 | 0
  Anxiety/depression, extremely anxious/depressed at BL | 0 | 0 | 1 | 0
  Anxiety/depression, not anxious/depressed at Week 12: number analyzed (Participants) | 5 | 6 | 5 | 1
  Anxiety/depression, not anxious/depressed at Week 12 | 4 | 2 | 4 | 1
  Anxiety/depression, moderately anxious/depressed at Week 12: number analyzed (Participants) | 5 | 6 | 5 | 1
  Anxiety/depression, moderately anxious/depressed at Week 12 | 1 | 4 | 1 | 0
  Anxiety/depression, extremely anxious/depressed at Week 12: number analyzed (Participants) | 5 | 6 | 5 | 1
  Anxiety/depression, extremely anxious/depressed at Week 12 | 0 | 0 | 0 | 0
  Anxiety/depression, not anxious/depressed at EOT: number analyzed (Participants) | 0 | 1 | 0 | 1
  Anxiety/depression, not anxious/depressed at EOT | 0 | 0 | 0 | 1
  Anxiety/depression, moderately anxious/depressed at EOT: number analyzed (Participants) | 0 | 1 | 0 | 1
  Anxiety/depression, moderately anxious/depressed at EOT | 0 | 1 | 0 | 0
  Anxiety/depression, extremely anxious/depressed at EOT: number analyzed (Participants) | 0 | 1 | 0 | 1
  Anxiety/depression, extremely anxious/depressed at EOT | 0 | 0 | 0 | 0

14. Secondary Outcome: Phase 2: Number of Participants With the Indicated Responses on the EQ-5D-3L Questionnaire Regarding Their Health State
Description: The EQ-5D-3L essentially consists of 2 components: the EQ-5D descriptive scale and the EQ-VAS. The EQ-5D-3L descriptive system comprises the following 5 dimensions: mobility, self-care, usual activities, anxiety/depression, and pain/discomfort. Each dimension has 3 levels: no problems, some problems, and extreme problems. At each specific visit (starting on Day 1), the participant was asked to indicate their health state.
Time Frame: up to 24 months
Population: as for outcome 4
Arm/Group | Recommended Phase 2 Dose (RP2D)
Number analyzed (Participants) | 0

15. Secondary Outcome: Phase 1: Cmax of Itacitanib
Description: Cmax was defined as the maximum observed concentration of itacitanib.
Time Frame: pre-dose and 1, 2, and 5 hours post-dose on Day 1 (Baseline) and at Week 4
Population: Pharmacokinetic (PK)-Evaluable Population: all enrolled participants who received at least 1 dose of itacitinib and provided at least 1 post-dose PK sample. Data were analyzed by dose rather than by treatment arm because approximately one-third of the participants had a dose adjustment (dose reduction) during the course of the study.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomoles per liter (nmol/L)
Groups:
- Itacitinib 200 mg QD: Participants received itacitinib 200 mg QD during the course of the study. Participants may have had dose reductions or modifications during the course of treatment based on adverse events, clinical evaluation, changes to concomitant medications, and laboratory assessments. Itacitinib treatment was continued until progression of bronchiolitis obliterans syndrome (defined as a ≥10% absolute decrease from Baseline in forced expiratory volume in 1 second (FEV1), confirmed by 2 consecutive spirometric assessments ≥3 weeks apart), unacceptable toxicity, loss of clinical benefit, or withdrawal of consent.
- Itacitinib 300 mg QD: Participants received itacitinib 300 mg QD during the course of the study. Participants may have had dose reductions or modifications during the course of treatment based on adverse events, clinical evaluation, changes to concomitant medications, and laboratory assessments. Itacitinib treatment was continued until progression of bronchiolitis obliterans syndrome (defined as a ≥10% absolute decrease from Baseline in forced expiratory volume in 1 second (FEV1), confirmed by 2 consecutive spirometric assessments ≥3 weeks apart), unacceptable toxicity, loss of clinical benefit, or withdrawal of consent.
- Itacitinib 300 mg BID: Participants received itacitinib 300 mg BID during the course of the study. Participants may have had dose reductions or modifications during the course of treatment based on adverse events, clinical evaluation, changes to concomitant medications, and laboratory assessments. Itacitinib treatment was continued until progression of bronchiolitis obliterans syndrome (defined as a ≥10% absolute decrease from Baseline in forced expiratory volume in 1 second (FEV1), confirmed by 2 consecutive spirometric assessments ≥3 weeks apart), unacceptable toxicity, loss of clinical benefit, or withdrawal of consent.
- Itacitinib 400 mg QD: Participants received itacitinib 400 mg QD during the course of the study. Participants may have had dose reductions or modifications during the course of treatment based on adverse events, clinical evaluation, changes to concomitant medications, and laboratory assessments. Itacitinib treatment was continued until progression of bronchiolitis obliterans syndrome (defined as a ≥10% absolute decrease from Baseline in forced expiratory volume in 1 second (FEV1), confirmed by 2 consecutive spirometric assessments ≥3 weeks apart), unacceptable toxicity, loss of clinical benefit, or withdrawal of consent.
- Itacitininb 600 mg QD: Participants received itacitinib 600 mg QD during the course of the study. Participants may have had dose reductions or modifications during the course of treatment based on adverse events, clinical evaluation, changes to concomitant medications, and laboratory assessments. Itacitinib treatment was continued until progression of bronchiolitis obliterans syndrome (defined as a ≥10% absolute decrease from Baseline in forced expiratory volume in 1 second (FEV1), confirmed by 2 consecutive spirometric assessments ≥3 weeks apart), unacceptable toxicity, loss of clinical benefit, or withdrawal of consent.
Arm/Group | Itacitinib 200 mg QD | Itacitinib 300 mg QD | Itacitinib 300 mg BID | Itacitinib 400 mg QD | Itacitininb 600 mg QD
Number analyzed (Participants) | 1 | 1 | 6 | 6 | 6
nanomoles per liter (nmol/L) | 370 (NA) — Dispersion cannot be reported for a single participant. | 2820 (NA) — Dispersion cannot be reported for a single participant. | 1820 (33.9) | 2050 (53.0) | 2410 (61.7)

16. Secondary Outcome: Phase 2: Cmax of Itacitanib
Description: Cmax was defined as the maximum observed concentration of itacitanib.
Time Frame: pre-dose and 1, 2, and 5 hours post-dose at Week 4
Population: as for outcome 4
Arm/Group | Recommended Phase 2 Dose (RP2D)
Number analyzed (Participants) | 0

17. Secondary Outcome: Phase 1: AUC0-24h of Itacitanib
Description: AUC0-24h was defined as the area under the plasma concentration-time curve over the last 24-hour dosing interval.
Time Frame: pre-dose and 1, 2, and 5 hours post-dose on Day 1 (Baseline) and at Week 4
Population: PK-Evaluable Population. Data were analyzed by dose rather than by treatment arm because approximately one-third of the participants had a dose adjustment (dose reduction) during the course of the study.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours x nmol/L
Arm/Group | Itacitinib 200 mg QD | Itacitinib 300 mg QD | Itacitinib 300 mg BID | Itacitinib 400 mg QD | Itacitininb 600 mg QD
Number analyzed (Participants) | 1 | 1 | 5 | 6 | 6
hours x nmol/L | 2590 (NA) — Dispersion cannot be reported for a single participant. | 33100 (NA) — Dispersion cannot be reported for a single participant. | 26800 (62.0) | 11900 (68.6) | 14300 (77.2)

18. Secondary Outcome: Phase 2: AUC0-24h of Itacitanib
Description: AUC0-24h was defined as the area under the plasma concentration-time curve over the last 24-hour dosing interval.
Time Frame: pre-dose and 1, 2, and 5 hours post-dose at Week 4
Population: as for outcome 4
Arm/Group | Recommended Phase 2 Dose (RP2D)
Number analyzed (Participants) | 0

19. Secondary Outcome: Phase 1: Tmax of Itacitanib
Description: tmax was defined as the time to the maximum observed concentration of itacitanib.
Time Frame: pre-dose and 1, 2, and 5 hours post-dose on Day 1 (Baseline) and at Week 4
Population: as for outcome 17
Measure: Median (Full Range); unit: hours
Arm/Group | Itacitinib 200 mg QD | Itacitinib 300 mg QD | Itacitinib 300 mg BID | Itacitinib 400 mg QD | Itacitininb 600 mg QD
Number analyzed (Participants) | 1 | 1 | 6 | 6 | 6
hours | 2.15 [NA to NA] — Full range cannot be reported for a single participant. | 4.63 [NA to NA] — Full range cannot be reported for a single participant. | 3.2 [1.8 to 4.5] | 2.0 [1.8 to 4.1] | 1.9 [1.0 to 4.0]

20. Secondary Outcome: Phase 2: Tmax of Itacitanib
Description: tmax was defined as the time to the maximum observed concentration of itacitanib.
Time Frame: pre-dose and 1, 2, and 5 hours post-dose at Week 4
Population: as for outcome 4
Arm/Group | Recommended Phase 2 Dose (RP2D)
Number analyzed (Participants) | 0

21. Secondary Outcome: Phase 1: Ctau of Itacitanib
Description: Ctau was defined as the observed itacitanib concentration at the end of the dosing interval.
Time Frame: pre-dose and 1, 2, and 5 hours post-dose on Day 1 (Baseline) and at Week 4
Population: as for outcome 17
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Arm/Group | Itacitinib 200 mg QD | Itacitinib 300 mg QD | Itacitinib 300 mg BID | Itacitinib 400 mg QD | Itacitininb 600 mg QD
Number analyzed (Participants) | 1 | 1 | 5 | 6 | 6
nmol/L | 9.34 (NA) — Dispersion cannot be reported for a single participant. | 403 (NA) — Dispersion cannot be reported for a single participant. | 510 (130) | 16.5 (675) | 43.4 (92.7)

22. Secondary Outcome: Phase 2: Ctau of Itacitanib
Description: Ctau was defined as the observed itacitanib concentration at the end of the dosing interval.
Time Frame: pre-dose and 1, 2, and 5 hours post-dose at Week 4
Population: as for outcome 4
Arm/Group | Recommended Phase 2 Dose (RP2D)
Number analyzed (Participants) | 0

23. Secondary Outcome: Phase 2: Time to Retransplantation or Death
Description: Time to retransplantation or death was defined as the interval between the start of treatment and the date of retransplantation or death due to any cause.
Time Frame: up to 24 months
Population: as for outcome 4
Arm/Group | Recommended Phase 2 Dose (RP2D)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: from the time of Informed Consent Form signing until at least 30 days after the last dose of study drug (up to approximately 3.67 years)
Description: Adverse events had been reported for members of the Full Analysis Set, comprised of all participants enrolled in the study who received at least 1 dose of itacitinib.
Arm/Group | Itacitinib 300/200 mg | Itacitinib 400/300 mg | Itacitinib 600/400 mg | Other
All-Cause Mortality (participants affected / at risk) | 0/7 | 2/7 | 2/8 | 0/1
Serious Adverse Events (participants affected / at risk) | 6/7 | 7/7 | 6/8 | 1/1
Other Adverse Events (participants affected / at risk) | 6/7 | 7/7 | 7/8 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Itacitinib 300/200 mg (N=7) | Itacitinib 400/300 mg (N=7) | Itacitinib 600/400 mg (N=8) | Other (N=1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acidosis hyperchloraemic (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 1 (2) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Bronchopulmonary aspergillosis (Infections and infestations) | 0 (0) | 2 (2) | 3 (3) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 3 (4) | 0 (0) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Cardiac death (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure acute (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cryptococcus test positive (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cytomegalovirus viraemia (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Donor specific antibody present (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
End stage renal disease (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Escherichia bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Herpes simplex pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Klebsiella bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Large intestine infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Metastatic squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myelodysplastic syndrome with single lineage dysplasia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Parainfluenzae virus infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia cytomegaloviral (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Pneumonia fungal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia pseudomonal (Infections and infestations) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Pneumonia viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pseudomonal bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Q fever (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Spinal synovial cyst (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Staphylococcal bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Systemic inflammatory response syndrome (General disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Transplant rejection (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tubulointerstitial nephritis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Itacitinib 300/200 mg (N=7) | Itacitinib 400/300 mg (N=7) | Itacitinib 600/400 mg (N=8) | Other (N=1)
Abdominal discomfort (Gastrointestinal disorders) | 2 (2) | 0 (0) | 2 (3) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 2 (3) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 2 (7) | 0 (0) | 0 (0)
Anaemia macrocytic (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Animal bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anogenital warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (4) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 2 (2) | 1 (2) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood cholesterol increased (Investigations) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Blood pressure increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (2) | 0 (0)
COVID-19 (Infections and infestations) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Cardiac flutter (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chest discomfort (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Colorectal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Congenital dyskeratosis (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Cushingoid (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cytomegalovirus infection reactivation (Infections and infestations) | 3 (4) | 3 (7) | 0 (0) | 0 (0)
Cytomegalovirus viraemia (Infections and infestations) | 2 (2) | 0 (0) | 2 (3) | 0 (0)
Deafness (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Defaecation urgency (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dental caries (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (2) | 1 (1) | 4 (5) | 0 (0)
Disseminated superficial actinic porokeratosis (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (2) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
End stage renal disease (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Enlarged uvula (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eye pain (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Fatigue (General disorders) | 2 (2) | 3 (3) | 3 (3) | 0 (0)
Feeling jittery (General disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Fluid retention (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastritis erosive (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Genital herpes (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gingival bleeding (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gout (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HCoV-OC43 infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3) | 1 (2) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 1 (8) | 2 (2) | 0 (0)
Herpes simplex (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Herpes simplex reactivation (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Herpes virus infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 2 (4) | 1 (1) | 0 (0)
Human polyomavirus infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 2 (2) | 3 (4) | 2 (2) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 2 (4) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Immunisation reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Immunosuppressant drug level increased (Investigations) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Iron deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 3 (4) | 1 (1) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lower respiratory tract infection bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Malaise (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Morganella infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myelocyte count increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nail discolouration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 2 (6) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ocular hypertension (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 3 (4) | 1 (1) | 0 (0)
Oesophageal candidiasis (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Onychomycosis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oral pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 2 (4) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Otitis externa (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Parainfluenzae virus infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Periorbital oedema (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peripheral swelling (General disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia pseudomonal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Polyp (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Prostatic specific antigen increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rectal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory syncytial virus infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory tract infection viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Retinal vein occlusion (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Right ventricular failure (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Scrotal pain (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Scrotal swelling (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Sjogren's syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0) | 0 (0) | 1 (1)
Sunburn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tendon disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (3) | 1 (1) | 1 (1) | 0 (0)
Tinea infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tinea versicolour (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Tongue disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tooth fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Transplant rejection (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Troponin increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection enterococcal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vasomotor rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 1 (4) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
A business decision was made to terminate the study before the initiation of Part 2. The decision to terminate the study was unrelated to safety concerns. Results from Phase 1 of the study have been reported in this summary.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Following the first publication, the Institution and/or Principal Investigator may publish data or results from the Study, provided, however, that the Institution and/or Principal Investigator submits the proposed publication to the Sponsor for review at least sixty (60) days prior to the date of the proposed publication. Sponsor may remove from the proposed publication any information that is considered confidential and/or proprietary other than Study data and results.

DOCUMENTS (2):
  • Study Protocol (2021-11-30): https://cdn.clinicaltrials.gov/large-docs/37/NCT03978637/Prot_000.pdf
  • Statistical Analysis Plan (2024-08-26): https://cdn.clinicaltrials.gov/large-docs/37/NCT03978637/SAP_001.pdf